CLINICAL TRIAL: NCT00658385
Title: A Pilot Trial to Assess the Feasibility and Safety of GCSF Mobilization of CD34+ Hematopoietic Progenitor Cells in Patients With Betathalassemia Major
Brief Title: Assess the Feasibility and Safety of Granulocyte Colony Stimulating Factor (GCSF) Mobilization of CD34+ Hematopoietic Progenitor Cells in Patients With Betathalassemia Major
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-030
Record Dates: First submitted 2008-04-10; First posted 2008-04-15 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Beta Thalassemia Major; Congenital Anemias
Keywords: GCSF
MeSH Terms: conditions — beta-Thalassemia | interventions — Leukapheresis

ARMS (1):
- 1 (Experimental): GCSF (human recombinant granulocyte colony stimulating factor)Neupogen(Amgen), Filgrastim, Central venous line placement, Stem cell Collection (leukapheresis)
  Interventions: Genetic: GCSF, Central venous line placement, Stem cell Collection (leukapheresis)

INTERVENTIONS:
Genetic: GCSF, Central venous line placement, Stem cell Collection (leukapheresis) — Daily injections under the skin of a GCSF. This is done for 5 to 6 days. On days 1, 3,5, and if need on day 6. To collect stem cells, we need good access to this blood. If the patient has good veins, we do this by placing an IV on each one of their arms. The peripheral blood stem cell collection is usually an outpatient procedure and takes about 3 to 4 hours. You will have blood work and a physical exam on days one, three, and five while you are getting GCSF.
  These will be done again 24 hours after your stem cells are collected.

SUMMARY:
Betathalassemia major is a disease of the blood and bone marrow. You were born with it and it has made you unable to make normal hemoglobin and red cells. You have been receiving red blood cell transfusions all your life. These transfusions do not cure your disease. The problem with transfusions is that they contain a lot of iron. With time iron builds up in your body and will eventually hurt some of your organs . Because of this buildup of iron , you are taking medicine that helps your body get rid of the extra iron.

Today, the only other treatment is bone marrow or stem cell transplant. It can only be done when a matched donor is available. This is most often a brother, sister, or parent. Bone marrow transplant may cure betathalassemia major. If you have a transplant and it is successful, you will no longer have the disease. Without a matched sibling or parent, the standard treatment is to keep having transfusions.

In the near future, we will be testing a new treatment for making normal hemoglobin and normal red blood cells. We have recreated the healthy hemoglobin gene in a test tube. We are able to use it and put it back into cells. This is called gene therapy. We have been able to put this gene into the stem cells of mice with thalassemia. These mice were cured. We now plan to take that gene and put it into stem cells from people who have betathalassemia major. We will then inject those stem cells back into that person's blood.

In general, we can obtain more stem cells from the blood of a person than from the bone marrow . In order to do so, we must give that person a blood growth factor. The growth factor stimulates the bone marrow to make more stem cells. That growth factor is called granulocyte colony stimulating factor (GCSF), or Filgrastim.

The purpose of this trial is to find out if the drug GCSF has any side effects on you, and if you will make more stem cells in response to it. This trial is not a gene therapy trial. This trial will not help your thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years or older
* Subjects may be of either gender or of any ethnic background
* Subjects must have a confirmed diagnosis of ßthalassemia major and have been enrolled in a hypertransfusion program with a confirmed annual transfusion of ≥ or = to 100 mL/kg/yr AND ≥ or = to 8 Transfusions of blood per year over a minimum of two years.
* Patients must be off hydroxyurea (HU) or erythropoietin (EPO) treatment for at least three months prior to entry onto the study
* Subjects must have a performance score of Karnofsky > or = to 70 of the time of entry into the study.
* Subjects must have a normal EKG and a normal chest xray
* Each patient must be willing to participate as a research subject and must sign an informed consent form.
* Subjects must be splenectomized or have no palpable spleen
* Negative pregnancy test, if female

Exclusion Criteria:

* Active infections including Hepatitis B and C, HTLV 1 and 2, West Nile Virus, and HIV 1
* Female patient pregnant or breast feeding
* Patients with uncontrolled seizure disorders
* Allergy to GCSF or bacterial E. coli products
* History of sickle cell disease or sickle trait
* History of thrombosis or known thrombophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farid Boulad, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- GCSF, Neupogen, Filgrastim, Central Venous Line Placement, SCT: GCSF (human recombinant granulocyte colony stimulating factor)Neupogen(Amgen), Filgrastim, Central venous line placement, Stem cell Collection (leukapheresis)
  GCSF, Central venous line placement, Stem cell Collection (leukapheresis): Daily injections under the skin of a GCSF. This is done for 5 to 6 days. On days 1, 3,5, and if need on day 6. To collect stem cells, we need good access to this blood. If the patient has good veins, we do this by placing an IV on each one of their arms. The peripheral blood stem cell collection is usually an outpatient procedure and takes about 3 to 4 hours. You will have blood work and a physical exam on days one, three, and five while you are getting GCSF.
  These will be done again 24 hours after your stem cells are collected.
Period: Overall Study
Arm/Group | GCSF, Neupogen, Filgrastim, Central Venous Line Placement, SCT
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GCSF, Neupogen, Filgrastim, Central Venous Line Placement, SCT
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With no Serious Adverse Events
Description: The entered value represents the number of participants with the absence of serious adverse events. G-CSF mobilization will be considered safe if there are no more than 1 of 5 patients with SAEs
Time Frame: Up to 14 Days
Measure: Number; unit: participants
Arm/Group | GCSF, Neupogen, Filgrastim, Central Venous Line Placement, SCT
Number analyzed (Participants) | 5
participants | 5

ADVERSE EVENTS:
Arm/Group | GCSF, Neupogen, Filgrastim, Central Venous Line Placement, SCT
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GCSF, Neupogen, Filgrastim, Central Venous Line Placement, SCT (N=5)
Blood bilirubin increased (Investigations) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes